CLINICAL TRIAL: NCT05963178
Title: Effects of an Early Logopedic Management and Speech Therapy in Post-Thyroidectomy Central Compartment Syndrome
Brief Title: Speech Therapy and Functional Dysphonia After Thyroidectomy
Acronym: LSCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, LONGOBARDI YLENIA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5604
Record Dates: First submitted 2023-07-05; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Functional Dysphonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Experimental)
  Interventions: Behavioral: Pre-operative counselling

INTERVENTIONS:
Behavioral: Pre-operative counselling — A preoperative speech therapy counseling will be carried out the day before the Total Thyroidectomy with the aim of informing patients about the possible conditions of the immediate post-operative period. Therefore, indications of vocal hygiene and hydration standards will be simultaneously administered, to be implemented from the first post-operative day.
  Patients will undergo phoniatric follow-up in the immediate post-operative period, at 7 days, 1 month and 3 months post-operatively.
  Patients who, at follow-up checks, should present the symptoms of functional post-thyroidectomy syndrome will undergo a cycle of post-operative speech therapy of 8 sessions.
  Other Names: Early speech therapy

SUMMARY:
Following a thyroidectomy, voice and swallowing alterations, which more frequently would appear to be caused by lesions of the laryngeal nerve, may occur. But, voice and swallowing changes can also occur in the absence of lesions of the inferior laryngeal nerve or the external branch of the superior laryngeal nerve, defining a condition called central compartment syndrome or functional post-thyroidectomy syndrome. It has been demonstrated that, in the presence of the aforementioned syndrome, the quality of the voice undergoes a deterioration immediately after thyroidectomy surgery with a lowering of pitch.

The purpose of this study will be to verify the effects of early speech therapy, including pre-operative speech therapy counseling (during which the patient will be provided with indications to be implemented in the immediate post-operative period).

ELIGIBILITY:
Inclusion Criteria:

* awaiting Total Thyroidectomy surgery
* able to sign a written consent

Exclusion Criteria:

* Under the age of 21 or over the age of 65
* Previous vocal cord paralysis
* History of vocal or laryngeal pathologies that have required therapy
* Presence of speech disorders or lung pathologies
* Previous neck surgery
* Presence of malignant diseases

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Acoustic analysis (f0) | 3 months
  Using the Multidimensional Voice Program, the Fundamental Frequency (F0, Hz) will be analyzed in the central 3 seconds of a sustained /a/.
Acoustic analysis (NHR) | 3 months
  Using the Multidimensional Voice Program, the noise/harmonics ratio (NHR) will be analyzed in the central 3 seconds of a sustained /a/.
Acoustic analysis (Jitter%) | 3 months
  Using the Multidimensional Voice Program, the Jitter (%) will be analyzed in the central 3 seconds of a sustained /a/.
Acoustic analysis (Shimmer%) | 3 months
  Using the Multidimensional Voice Program, the Shimmer (%) will be analyzed in the central 3 seconds of a sustained /a/.
Voice Range Profile (Flow) | 3 months
  The patient will be instructed in the production of a sustained /a/ from the lowest to the highest note, from minimum to maximum intensity. In this case, the Minimum frequency (Flow) will be analysed.
Voice Range Profile (Fhigh) | 3 months
  The patient will be instructed in the production of a sustained /a/ from the lowest to the highest note, from minimum to maximum intensity. In this case, the Maximum frequency (Fhigh) will be analysed.
Voice function | 3 months
  A questionnaire called Voice Impairment Score (VIS) will be used, created specifically to investigate the frequency of voice alterations. The VIS consists of 10 items and can vary from a minimum score of 0 (no vocal alteration) to a maximum of 40 (maximum voice disturbance).
Swallowing function | 3 months
  A questionnaire called Swallowing Impariment Scores (SIS) will be used, created specifically to investigate the frequency of swallowing alterations. The SIS consists of 5 items and can vary from a minimum score of 0 (no vocal alteration) to a maximum of 20 (maximum swallowing disturbance).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli - IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No